CLINICAL TRIAL: NCT05785975
Title: Effectiveness of Modified Integrated Colorectal Cancer Screening System: A Randomized Clustered Trial in Hail, Saudi Arabia.
Brief Title: Effectiveness of Modified Integrated Colorectal Cancer Screening System in Saudi Arabia
Acronym: ColonCancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The New Model of Care, Hail Health Cluster (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: New Model of Care Hail Cluster
Record Dates: First submitted 2023-02-27; First posted 2023-03-27 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention is an integrated system built on the concept of nudging and made up of a trained family doctor, community outreach (using landline calls, and a single FIT test for occult blood. Together with the information, education, and communication (IEC) texts that were sent to the outreach participants by SMS. four screening healthcare zones that included 34 public primary care facilities in the Hail region.
  The total sample size for the two trial arms is 2520 individuals. The calculation was done using the STATA version 15 data analysis software, the sample size command, and the cluster sizes of m1 = (60), m2 = (60), a control-group rate of (0.4), an experimental group rate of (0.6), the intraclass correlation coefficient (rho) of (0.02), a power beta of (0.8), and a sample of N1 = (1260), N2 = (1260).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Certain ommunications(Nudge), community-outreach(landline call), and single FIT testing (Experimental): The intervention is an integrated system made up of single FIT testing, community outreach (landline call), and specific messages (Nudge). In order to encourage people to attend the screening, a primary care physician will be used in addition to text messages that participants at the outreach get for information, education, and communication (IEC).
  Interventions: Other: Certain ommunications(Nudge), community-outreach(landline call), and single FIT testing
- Routine Care for colorectal cancer screening (No Intervention): The comparators will be individuals with an average risk of colorectal cancer of both genders attending the selected health centres / or recruited through a community outreach approach.

INTERVENTIONS:
Other: Certain ommunications(Nudge), community-outreach(landline call), and single FIT testing — The intervention is an integrated system made up of single FIT testing, community outreach (landline call), and specific messages (Nudge). In order to encourage people to attend the screening, a primary care physician will be used in addition to text messages that participants at the outreach get for information, education, and communication (IEC).
  Arms: Certain ommunications(Nudge), community-outreach(landline call), and single FIT testing

SUMMARY:
In order to encourage the population at risk to participate in colorectal cancer screening, this clustered trial intends to determine the efficacy of specific messages(Nudge), single FIT testing, and the primary care physician's clinical judgment on referral to colonoscopy.

It primarily seeks to provide answers to the following questions: How effective is the modified integrated CRC screening system (MICRCSS) for individuals with average colorectal cancer risk? based on the percentage of individuals who had CRC screening, registered for the follow-up, and were discovered to have precancerous CRC issues a year after the program's start, as contrasted to individuals receiving standard medical care? All public government entities in the Hail region will be contacted with invitations to participate in the study (outreach). the organization

DETAILED DESCRIPTION:
Introduction:

Incidence of colorectal cancer (CRC), which starts in the innermost lining mucosa of the colon or rectum, is third (10.2%) in the globe behind lung and breast cancers (11,6%), according to the Global Cancer Observatory (GCO) 2018. According to a 2010 research, Saudi Arabia had an incidence of 10.4/100,000; regrettably, the incidence among young age groups is greater than that in countries with high incidence.

The majority of colorectal malignancies (CRCs) are first identified as polyps, which are small benign growths or projections seen inside the lumen of the colon. If a polyp is larger than 1 cm, if there are more than two polyps present, or if dysplasia is seen after the polyp is removed, the polyp is considered to be precancerous. Precancerous adenomas, hyperplastic polyps, or inflammatory polyps

ELIGIBILITY:
Inclusion Criteria:

* Age 40 -75

Exclusion Criteria:

* Sever ill patient

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2520 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the CRC screening enrollment rates between the intervention and control groups. | 6 month from the start of the study
  The proportion of people who had CRC screening who were included in the intervention group as opposed to the control group
To assess if positive subjects are complying with follow-up screening | 6 month from the start of the study
  The proportion of participants in the intervention group compared to the control group who tested positive and underwent a colonoscopy as a follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Khalil I Alshammari, VIP Chief MO, Study Chair — Hail Health Cluster; Meshari Aljamaani, MOC Lead, Study Director — New Model of Care, Hail Health Cluser; Fakhralddin A Elfakki, Research Lead, Principal Investigator — New Model of Care, Hail Health Cluster
Locations (1):
- Al Hait General Hospital Zone, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The research outcome will be shared at the Saudi conference for pathway improvement
Supporting Information: CSR
Time Frame: September 2023
Access Criteria: Data will be available in August 2023

REFERENCES:
- [Derived] Elfakki FAM, Alshammari KI, Aljamani MY, Alshammari WI. A nudge strategy to increase the uptake of colorectal cancer screening in Saudi Arabia: A pragmatic randomized trial in the Hail region. J Family Med Prim Care. 2024 Jan;13(1):163-168. doi: 10.4103/jfmpc.jfmpc_966_23. Epub 2024 Feb 8. PMID 38482290